CLINICAL TRIAL: NCT01082029
Title: Role of Empiric Anti-reflux Therapy in Pediatric Otitis Media With Effusion - a Pilot Study
Brief Title: Study of Anti-reflux Medication as a Potential Treatment for Glue Ear in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Gavin Rukholm, Dr Gavin Rukholm, MD FRCSC, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-435
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lansoprazole (Experimental)
  Interventions: Drug: Lansoprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lansoprazole — The dosage of Lansoprazole will be administered based on guidelines set out by the prescription drug information outlined in the official Lansoprazole package insert and will remain the same for each patient during the 3 month period and is as follows: a) 1 to 11 years of age, weight less then or equal to 30 kg, 15 mg orally once daily. b) 1 to 11 years of age, weight greater then 30 kg, 30 mg orally once daily. c) 12 years of age and older, 15 mg orally once daily. The doses of Lansoprazole will be prepared in liquid form by the Inpatient Pharmacy at Hamilton Health Sciences.
  Other Names: Prevacid
  Arms: Lansoprazole
Drug: Placebo — Lactose powder in 8.4% Sodium Bicarbonate (Liquid placebo)
  Arms: Placebo

SUMMARY:
The accumulation of fluid behind the ear drum without any acute inflammation is known as otitis media with effusion (OME). It is the most common cause of acquired hearing loss during childhood. Long-term complications of OME include linguistic, developmental, and social development delays due to hearing loss.

The cause of OME is not known; however, low grade infection of the middle ear, poor function of the eustachian tube between the ear and the throat, and adenoid hypertrophy have all been suggested as possible etiologies. Recent detection of the stomach enzyme pepsin in middle ear fluid has led some to propose that OME is related to the reflux of stomach contents into the ear, via the eustachian tube.

The purpose of the investigators study is to determine whether anti-reflux medication may have a positive impact by clearing the accumulation of fluid in the middle ear with the aim of preventing or reducing hearing loss in children diagnosed with OME. Empiric anti-reflux therapy with proton pump inhibitor (PPI) medication is safe, proven and cost-effective. It is used widely as a diagnostic and treatment strategy in the presence of the signs and symptoms of gastroesophageal reflux disease (GERD). The signs and symptoms of GERD include heartburn, recurrent vomiting or regurgitation, acid taste in mouth, throat irritation, voice problems, heartburn, difficult or painful swallowing, asthma and recurrent pneumonia.

This pilot study will be a double-blinded, randomized, placebo-controlled trial that will compare resolution rates for OME in children treated with lansoprazole or placebo for three months. At the end of the study, those patients who have persistent middle ear effusions will be brought to the operating room and have the fluid aspirated and sent for analysis for pepsin.

DETAILED DESCRIPTION:
Otitis media with effusion (OME) is a condition characterized by the accumulation of non-purulent fluid in the middle ear space, in the absence of acute inflammation. OME is diagnosed 2.2 million times annually (U.S. Department of Health & Human Services, 2000). It is a condition in which more then 50% of children will experience in their first year of life (National Institutes of Health, 1993). Although many episodes resolve spontaneously, 30% to 40% persist, and 5% to 10% of episodes last 1 year or longer (Yoshinaga-Itano, 1995). It is particularly more common among children between the ages of one and three years and in seasons where the prevalence of upper respiratory tract infections is high; with an incidence of 10% to 30%. It occurs frequently even up to the age of seven, with a prevalence of 3% to 8%(Fiellau et al, 1997; Fiellau et al, 1983; Lous et al, 1981; Teele et al, 1989).

OME is the most common cause of acquired hearing loss in childhood. Long-term hearing complications from OME are associated with linguistic, developmental, and social consequences; especially if the OME is bilateral and of long duration (Fiellau et al, 1983; Golz et al, 1998; Grace et al, 1990; Lous et al, 1995). The etiology of OME is uncertain; however, low-grade infection, poor eustachian tube function, formation of biofilms, and adenoidal infection or hypertrophy have all been suggested as possible etiologies (Faden et al, 1998; Hall-Stoodley et al, 2006).

Recently, there has been good scientific evidence to suggest that OME is a supraesophageal manifestation of gastroesophageal reflux disease (GERD), and more specifically laryngo-pharyngeal reflux (LPR). Tasker et al (2002) investigated the potential role of gastric reflux in the development of OME in children who underwent myringotomy. Of 65 tested effusion samples, 59 (91%) effusions gave a positive result. The concentrations of pepsin/pepsinogen were roughly estimated to be about 1000 times higher than those found in the serum obtained from a number of controls. They speculated that pepsin found in middle ear effusion (MEE) was most probably due to micro-aspiration of gastric contents passing through the eustachian tube (ET) and reaching the middle ear. Lieu et al (2005) performed a pilot study where they replicated the finding of pepsin/pepsinogen in 17 of 36 (77%) middle ear fluid aspirates, obtained from 22 children who underwent tympanostomy tube placement for chronic or recurrent otitis media (OM).

Based on our literature review, we believe there is sufficient scientific evidence to support the empiric treatment of suspected GERD and LPR in patients with OME. Empiric anti-reflux therapy is a safe, proven, cost-effective diagnostic and treatment strategy used widely in the presence of other signs and symptoms of suspected GERD. This pilot study will be a double-blinded, randomized control trial. It will compare hearing outcomes for children with OME being treated with lansoprazole versus placebo for three months. We believe there is sufficient evidence to support the use of this strategy in patients with suspected GERD and LPR who present with OME.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 1 and 17 years referred to the McMaster Otolaryngology Clinic.
* Presence of bilateral OME for at least 3 months based on:

  * Clinical history: patient may present with decrease in hearing, aural fullness and/or ear pressure, balance problems, ear tugging/rubbing, they typically do not have otalgia or fever.
  * Pneumatic otoscopy: observations suggestive of OME include presence of a dull tympanic membrane with presence of non purulent effusion (serous or mucoid), presence of a level of effusion, decrease or non motility of the tympanic membrane, retraction of the tympanic membrane.
  * Tympanometry: type B or type C tympanogram with normal air volume of the external auditory canal.
  * Pure tone audiometry: conductive hearing loss that typically varies from slight to moderate.

Exclusion Criteria:

* Presence of acute otitis media as determined by history and physical examination:

  * History of rapid acute onset of significant otalgia, decrease in hearing, fever, irritability.
  * Pneumatic otoscopy revealing purulent effusion, yellowness and/or redness with hypervascularity of the tympanic membrane, bulging of tympanic membrane with decrease of normal landmarks.
* Presence of craniofacial abnormalities
* Previous middle ear surgery (excluding myringotomy and tube)
* Allergic reactions to lansoprazole, and any other adverse drug interactions to lansoprazole.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2010-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Collect the required data for sample size calculation | Following the recruitment of 100 patients (~1 year)
  The purpose of this pilot study is to collect required data for a sample size calculation for a larger clinical trial and to determine recruitment rates.

SECONDARY OUTCOMES:
Resolution of Otitis Media with Effusion | At presentation and at 1 month, 2months and 3 months post initiation of treatment
  The secondary objectives are to compare the duration of OME between the placebo and treatment groups, and to compare the duration and degree of hearing loss at initial presentation and at three months. Other outcomes include degree of hearing improvement, complications of OME (i.e. recurrent OME, acute otitis media, surgery), frequency and severity of GERD symptoms, side effects of Lansoprazole use, and presence of pepsin in middle ear effusions collected from patients who received surgical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Diane Reid, MD FRCSC, Principal Investigator — McMaster University; Dr. Gavin Rukholm, MD, Principal Investigator — McMaster University
Locations (1):
- Mcmaster University Medical Centre 3V1 Clinic, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Bluestone CD, Beery QC, Andrus WS. Mechanics of the Eustachian tube as it influences susceptibility to and persistence of middle ear effusions in children. Ann Otol Rhinol Laryngol. 1974 Mar-Apr;83:Suppl 11:27-34. doi: 10.1177/0003489474083s1103. No abstract available. PMID 4819098
- [Background] Charbel S, Khandwala F, Vaezi MF. The role of esophageal pH monitoring in symptomatic patients on PPI therapy. Am J Gastroenterol. 2005 Feb;100(2):283-9. doi: 10.1111/j.1572-0241.2005.41210.x. PMID 15667483
- [Background] Crapko M, Kerschner JE, Syring M, Johnston N. Role of extra-esophageal reflux in chronic otitis media with effusion. Laryngoscope. 2007 Aug;117(8):1419-23. doi: 10.1097/MLG.0b013e318064f177. PMID 17585281
- [Background] Deal L, Gold BD, Gremse DA, Winter HS, Peters SB, Fraga PD, Mack ME, Gaylord SM, Tolia V, Fitzgerald JF. Age-specific questionnaires distinguish GERD symptom frequency and severity in infants and young children: development and initial validation. J Pediatr Gastroenterol Nutr. 2005 Aug;41(2):178-85. doi: 10.1097/01.mpg.0000172885.77795.0f. PMID 16056096
- [Background] Fass R, Ofman JJ, Gralnek IM, Johnson C, Camargo E, Sampliner RE, Fennerty MB. Clinical and economic assessment of the omeprazole test in patients with symptoms suggestive of gastroesophageal reflux disease. Arch Intern Med. 1999 Oct 11;159(18):2161-8. doi: 10.1001/archinte.159.18.2161. PMID 10527293
- [Background] Fiellau-Nikolajsen M, Lous J, Vang Pedersen S, Schousboe HH. Tympanometry in three-year-old children. I. A regional prevalence study on the distribution of tympanometric results in a non-selected population of 3-year-old children. Scand Audiol. 1977;6(4):199-204. doi: 10.3109/01050397709043121. PMID 609889
- [Background] Fiellau-Nikolajsen M, Lous J. Prospective tympanometry in 3-year-old children. A study of the spontaneous course of tympanometry types in a nonselected population. Arch Otolaryngol. 1979 Aug;105(8):461-6. doi: 10.1001/archotol.1979.00790200023005. PMID 464883
- [Background] Fiellau-Nikolajsen M. Tympanometry and secretory otitis media. Observations on diagnosis, epidemiology, treatment, and prevention in prospective cohort studies of three-year-old children. Acta Otolaryngol Suppl. 1983;394:1-73. No abstract available. PMID 6314732
- [Background] Gerson LB, Robbins AS, Garber A, Hornberger J, Triadafilopoulos G. A cost-effectiveness analysis of prescribing strategies in the management of gastroesophageal reflux disease. Am J Gastroenterol. 2000 Feb;95(2):395-407. doi: 10.1111/j.1572-0241.2000.01759.x. PMID 10685741
- [Background] Golz A, Netzer A, Angel-Yeger B, Westerman ST, Gilbert LM, Joachims HZ. Effects of middle ear effusion on the vestibular system in children. Otolaryngol Head Neck Surg. 1998 Dec;119(6):695-9. doi: 10.1016/S0194-5998(98)70039-7. PMID 9852553
- [Background] Grace AR, Pfleiderer AG. Dysequilibrium and otitis media with effusion: what is the association? J Laryngol Otol. 1990 Sep;104(9):682-4. doi: 10.1017/s0022215100113611. PMID 2230572
- [Background] Heavner SB, Hardy SM, White DR, Prazma J, Pillsbury HC 3rd. Transient inflammation and dysfunction of the eustachian tube secondary to multiple exposures of simulated gastroesophageal refluxant. Ann Otol Rhinol Laryngol. 2001 Oct;110(10):928-34. doi: 10.1177/000348940111001007. PMID 11642425
- [Background] Hicks DM, Ours TM, Abelson TI, Vaezi MF, Richter JE. The prevalence of hypopharynx findings associated with gastroesophageal reflux in normal volunteers. J Voice. 2002 Dec;16(4):564-79. doi: 10.1016/s0892-1997(02)00132-7. PMID 12512644
- [Background] Jonaitis L, Pribuisiene R, Kupcinskas L, Uloza V. Laryngeal examination is superior to endoscopy in the diagnosis of the laryngopharyngeal form of gastroesophageal reflux disease. Scand J Gastroenterol. 2006 Feb;41(2):131-7. doi: 10.1080/00365520600577940. PMID 16484116
- [Background] Keles B, Ozturk K, Gunel E, Arbag H, Ozer B. Pharyngeal reflux in children with chronic otitis media with effusion. Acta Otolaryngol. 2004 Dec;124(10):1178-81. doi: 10.1080/00016480410017134. PMID 15768814
- [Background] Lieu JE, Muthappan PG, Uppaluri R. Association of reflux with otitis media in children. Otolaryngol Head Neck Surg. 2005 Sep;133(3):357-61. doi: 10.1016/j.otohns.2005.05.654. PMID 16143181
- [Background] Lous J, Fiellau-Nikolajsen M. Epidemiology and middle ear effusion and tubal dysfunction. A one-year prospective study comprising monthly tympanometry in 387 non-selected 7-year-old children. Int J Pediatr Otorhinolaryngol. 1981 Dec;3(4):303-17. doi: 10.1016/0165-5876(81)90055-0. PMID 6976949
- [Background] Lous J. Secretory otitis media in schoolchildren. Is screening for secretory otitis media advisable? Dan Med Bull. 1995 Feb;42(1):71-99. No abstract available. PMID 7729171
- [Background] Rodriguez-Tellez M. Supra-oesophageal manifestations of gastro-oesophageal reflux disease. Drugs. 2005;65 Suppl 1:67-73. doi: 10.2165/00003495-200565001-00010. PMID 16335860
- [Background] Rozmanic V, Velepic M, Ahel V, Bonifacic D, Velepic M. Prolonged esophageal pH monitoring in the evaluation of gastroesophageal reflux in children with chronic tubotympanal disorders. J Pediatr Gastroenterol Nutr. 2002 Mar;34(3):278-80. doi: 10.1097/00005176-200203000-00009. PMID 11964951
- [Background] Shekelle P, Takata G, et al. Diagnosis, Natural History, and Late Effects of Otitis Media with Effusion. Evidence Report/Technology Assessment No. 55 (Prepared by Southern California Evidence-based Practice Center under Contract No 290-97-0001, Task Order No. 4). AHRQ Publication No. 03-E023. Rockville, MD: Agency for Healthcare Research and Quality May 2003.
- [Background] Tasker A, Dettmar PW, Panetti M, Koufman JA, P Birchall J, Pearson JP. Is gastric reflux a cause of otitis media with effusion in children? Laryngoscope. 2002 Nov;112(11):1930-4. doi: 10.1097/00005537-200211000-00004. PMID 12439157
- [Background] Teele DW, Klein JO, Rosner B. Epidemiology of otitis media during the first seven years of life in children in greater Boston: a prospective, cohort study. J Infect Dis. 1989 Jul;160(1):83-94. doi: 10.1093/infdis/160.1.83. PMID 2732519
- [Background] White DR, Heavner SB, Hardy SM, Prazma J. Gastroesophageal reflux and eustachian tube dysfunction in an animal model. Laryngoscope. 2002 Jun;112(6):955-61. doi: 10.1097/00005537-200206000-00004. PMID 12160291
- [Background] Vaezi MF. Therapy Insight: gastroesophageal reflux disease and laryngopharyngeal reflux. Nat Clin Pract Gastroenterol Hepatol. 2005 Dec;2(12):595-603. doi: 10.1038/ncpgasthep0358. PMID 16327839
- [Background] Velepic MM, Velepic MS, Starcevic R, Manestar D, Rozmanic V. Gastroesophageal reflux and sequelae of chronic tubotympanal disorders in children. Acta Otolaryngol. 2004 Oct;124(8):914-7. doi: 10.1080/00016480410022499. PMID 15513526
- [Background] Al-Saab F, Manoukian JJ, Al-Sabah B, Almot S, Nguyen LH, Tewfik TL, Daniel SJ, Schloss MD, Hamid QA. Linking laryngopharyngeal reflux to otitis media with effusion: pepsinogen study of adenoid tissue and middle ear fluid. J Otolaryngol Head Neck Surg. 2008 Aug;37(4):565-71. PMID 19128594